CLINICAL TRIAL: NCT00627588
Title: A Phase I/II Study of the Safety, Efficacy and Dose Evaluation of ProSavin®, Administered Using Stereotactic Injection to the Striatum of Patients With Bilateral, Idiopathic Parkinson's Disease.
Brief Title: Phase I/II Study of the Safety, Efficacy and Dose Evaluation of ProSavin for the Treatment of Bilateral Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oxford BioMedica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS-001-07; EudraCT Number: 2007-001109-26
Record Dates: First submitted 2008-01-31; First posted 2008-03-03 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Parkinson's Disease
Keywords: ProSavin; Parkinson's Disease; Gene Therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose Evaluation (Experimental): To assess the safety and efficacy of up to three dose levels of ProSavin
  Interventions: Biological: ProSavin
- Sham element (Sham Comparator): The potential use of sham comparator to confirm efficacy
  Interventions: Biological: ProSavin

INTERVENTIONS:
Biological: ProSavin — ProSavin is a gene therapy designed to delivery three key enzymes involved in the synthesis of dopamine
  Arms: Dose Evaluation
Biological: ProSavin — ProSavin is a gene therapy designed to delivery three key enzymes involved in the synthesis of dopamine
  Arms: Sham element

SUMMARY:
The primary objectives of the trial are to assess the safety and efficacy of ProSavin.

Patients in the trial will have been diagnosed with Parkinson's disease and will be failing on current treatment with L-DOPA but they will not have progressed to drug-induced dyskinesias. The first stage is an open-label dose escalation to evaluate up to three dose levels of ProSavin in cohorts of three patients each. Following a recommendation by the DMC the study may proceed to the second stage of the trial, a further 12 patients will be recruited to confirm efficacy of the optimal dose in the randomized phase of the study.

The efficacy of ProSavin will be assessed using the Unified Parkinson's Disease Rating Score (UPDRS). Patients will be monitored at regular intervals, with the primary endpoint being an efficacy assessment at six months after treatment. The secondary objective of the trial is to asses the extent to which patients' current therapy (L-DOPA) can be reduced following administration of ProSavin.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written Informed Consent
2. Diagnosed with bilateral idiopathic PD
3. Diagnosis of PD > five years, using diagnostic criteria from core assessment program for surgical interventional therapies CAPSIT (1999)
4. Males/females between 48 and 65 years
5. Women must be postmenopausal, with last menstrual period being over two years ago
6. Male patients must agree to use at least two methods of contraception for at least 3 months following ProSavin administration if they and their partner is of child-bearing capacity
7. Response to L-DOPA where an increase in dose is unacceptable to the patient due to potentiating the fluctuations in motor functions
8. Hoehn and Yahr stage 3 and 4
9. UPDRS (Part III) of between 20 and 60 in the "OFF" state
10. Stable dosing of PD medication, including L-DOPA, for six weeks prior to surgery
11. Positive response to dopaminergic therapy as defined by a 50% improvement in UPDRS (Part III) between the "OFF" and "ON" states
12. Presence of motor fluctuations
13. Willing to have current treatment withdrawn for up to 24 hours prior to surgery therefore being in an "OFF" state for surgery
14. Willing to have their L-DOPA dosage reduced/withdrawn at the discretion of the principal investigator (PI) at regular intervals following surgery to allow assessment of ProSavin in the absence of concomitant anti-{Parkinsonian medication
15. Affiliated with the French social security health care system (Patients enrolled in France only)

Exclusion Criteria:

1. Major surgery within the 28 days prior to enrolment
2. Severe disabling dyskinesias > or = 51% of the day as defined by the UPDRS (Part IV)
3. History of psychosis or current treatment with dopamine blocking agents of any kind
4. Severe depression as defined by a BDI score of >16. Any treatment for depression should be limited to seretonergic therapies and those that do not target the dopaminergic pathways
5. Prior treatment with tolcapone within the six months prior to enrollment into the study, due to its ability to modify dopaminergic pathways in the brain
6. History of epilepsy or any other co-morbid condition that the Investigator believes presents an unacceptable health risk to the patient in conjunction with the procedures in this protocol
7. Life-threatening illness unrelated to PD
8. History of stereotactic or other surgery for the treatment of PD
9. Premenopausal women
10. Alcohol or other substance abuse
11. Clinically significant laboratory test abnormalities, including full blood count, chemistry panel, liver function tests, electrocardiogram (ECG), Chest X rays
12. Any contraindication for undergoing an MRI scan of the head
13. Intercurrent illness or infection 28 days prior to enrolment
14. Abnormal MRI findings such as mega cisterna, septum pellucidum, signs of severe cortical or subcortical atrophy, brain tumours, vascular diseases, trauma or arteriovenous malformations (AVM)
15. Prior regular exposure to neuroleptic agents
16. History of treatment with any agent that may induce PD or PD symptoms within the last three months prior to enrollment
17. Contraindications to use of anaesthesia
18. Treated with dopaminergic antagonists six months prior to screening
19. Concurrent antiretroviral therapy that would inactivate the investigational agent
20. History of any investigational agent within 28 days prior to ProSavin administration
21. Participation in a prior gene transfer therapy study
22. Enrolment in any other clinical study, for any condition, including those relating to PD, throughout the duration of the ProSavin study
23. Current of anticipated treatment with anticoagulant therapy or the use of anticoagulation therapy within the four weeks prior to surgery
24. Diagnosis of multiple systems atrophy (MSA) following assessment of the autonomic nervous systems function (e.g. blood pressure, difficulty in urinating and sexual activity) and MRI during the screening process
25. Administration of subcutaneous rescue remedy apomorphine
26. Patient unable to adhere to their prescribed Parkinson's disease treatment regime.

Ages: 48 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Safety as measured by the number and severity of Adverse Events | 1 year

SECONDARY OUTCOMES:
Efficacy as measured by the UPDRS | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Palfi, Professor, Principal Investigator — Henri Mondor University Hospital
Locations (2):
- Henri Mondor Hospital, Paris, France
- Addenbrookes Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Palfi S, Gurruchaga JM, Ralph GS, Lepetit H, Lavisse S, Buttery PC, Watts C, Miskin J, Kelleher M, Deeley S, Iwamuro H, Lefaucheur JP, Thiriez C, Fenelon G, Lucas C, Brugieres P, Gabriel I, Abhay K, Drouot X, Tani N, Kas A, Ghaleh B, Le Corvoisier P, Dolphin P, Breen DP, Mason S, Guzman NV, Mazarakis ND, Radcliffe PA, Harrop R, Kingsman SM, Rascol O, Naylor S, Barker RA, Hantraye P, Remy P, Cesaro P, Mitrophanous KA. Long-term safety and tolerability of ProSavin, a lentiviral vector-based gene therapy for Parkinson's disease: a dose escalation, open-label, phase 1/2 trial. Lancet. 2014 Mar 29;383(9923):1138-46. doi: 10.1016/S0140-6736(13)61939-X. Epub 2014 Jan 10. PMID 24412048